CLINICAL TRIAL: NCT00481741
Title: A Prospective Randomized Controlled Efficacy and Safety Trial of the SafeSeal Hemostasis Patch Compared to Manual Compression for Achieving Vascular Hemostasis Following Percutaneous Coronary and Peripheral Intervention.
Brief Title: Study of the SafeSeal(TM) Hemostasis Patch Following Percutaneous Coronary Artery and Peripheral Vascular Interventions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: MEDRAD, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00018198
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Coronary Artery Disease; Peripheral Vascular Disease
Keywords: Angioplasty, Percutaneous TransluminalCoronary
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SafeSeal(TM) Hemostasis Patch

SUMMARY:
We seek to determine if the use of the SafeSeal(TM) topical hemostasis patch is associated with reductions in time to hemostasis and time to ambulation compared to standard manual compression after arterial sheath removal following percutaneous coronary and peripheral intervention. We further seek to assess the safety of the SafeSeal patch compared to manual compression.

DETAILED DESCRIPTION:
A variety of topical hemostasis pads containing procoagulant materials are currently available to accelerate hemostasis after removal of the arterial introducer sheath following coronary and peripheral arterial angioplasty procedures. The effectiveness and safety of these pads, however, remains poorly understood. A total of 150 patients undergoing coronary or peripheral vascular angioplasty through a 6 French arterial sheath will be randomized to sheath removal using manual compression alone or manual compression combined with use of the SafeSeal(TM) hemostasis patch. Sheaths will be removed at an activated clotting time (ACT) of <250 seconds, and patients will be kept at bedrest for 2 hours after hemostasis is achieved. The primary endpoint will be time to hemostasis. Secondary endpoints witll include time to ambulation and frequency of bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old
2. Coronary or peripheral vascular intervention
3. 6 French arterial sheath used
4. Overnight hospitalization following procedure

Exclusion Criteria:

1. Hematoma or persistent bleeding around the vascular sheath
2. Previous AV fistula or pseudoaneurysm in the ipsilateral femoral artery
3. History of bleeding diathesis or coagulopathy
4. Hemoglobin level < 9 g/dl
5. Inability to ambulate at baseline
6. Known allergy to any of the materials used in the SafeSeal
7. Female patients known to be pregnant or lactating
8. Evidence of ongoing systemic or cutaneous infection
9. Uncontrolled blood pressure following PCI (systolic blood pressure > 180 or diastolic blood pressure >110)
10. Current enrolment in another ongoing investigational drug/device trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to achieve hemostasis of femoral artery after arterial sheath removal | immediate

SECONDARY OUTCOMES:
vascular access-related bleeding complications | prior to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Narins, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States